CLINICAL TRIAL: NCT04968613
Title: Dopaminergic Mechanism of Temporal Working Memory Impairment in Parkinson's Disease
Brief Title: Dopaminergic Mechanism of Memory Impairment in Parkinson's Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Chinese Academy of Sciences (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: M2017368
Record Dates: First submitted 2021-06-27; First posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-06

CONDITIONS: Parkinson Disease; Memory Impairment
MeSH Terms: conditions — Parkinson Disease; Memory Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Madopar monotherapy group (Experimental): Patients in this group received Madopar monotherapy
  Interventions: Drug: Madopar monotherapy
- senfrol monotherapy group (Active Comparator): Patients in this group were treated with senfrol (D2 receptor agonist) alone
  Interventions: Drug: senfrol monotherapy
- placebo group (Placebo Comparator): Patients in this group were treated with selegiline alone
  Interventions: Drug: placebo monotherapy

INTERVENTIONS:
Drug: Madopar monotherapy — In addition to basic treatment, the patient also received Madopar treatment
  Arms: Madopar monotherapy group
Drug: senfrol monotherapy — In addition to the basic treatment, the patient also received the rofosson treatment
  Arms: senfrol monotherapy group
Drug: placebo monotherapy — In addition to basic treatment, the patient also received selegiline treatment
  Arms: placebo group

SUMMARY:
The cognitive impairment of Parkinson's disease is non amnestic, which is characterized by working memory impairment and executive dysfunction. The current drug therapy (such as levodopa, dopamine receptor agonists) and surgical treatment (such as deep brain electrical stimulation, thalamic lesion) not only can not effectively alleviate cognitive impairment, but also may aggravate cognitive and speech behavior abnormalities. This project will explore how dopamine regulates temporal working memory in human research by combining drug intervention, neuroimaging and cognitive tasks.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a common neurodegenerative disease in the elderly. The incidence rate of China's disease is 1.7% in the population over 65 years old. The latest research shows that Parkinson's disease is not a simple motor disorder, but a multi organ dysfunction disorder with both motor symptoms and non motor symptoms. With the development of the disease, more than 80% of the PD patients will develop dementia. Different from the amnestic cognitive impairment of Alzheimer's disease, the cognitive impairment of Parkinson's disease is non amnestic, characterized by working memory impairment and executive dysfunction. The current mainstream drug therapy (such as levodopa, dopamine receptor agonists) and surgical treatment (such as deep brain electrical stimulation, thalamic lesion) can not effectively alleviate cognitive impairment, and may even aggravate cognitive and speech behavior abnormalities, We should first understand the neurochemical (molecular) mechanisms of working memory impairment and executive dysfunction in Parkinson's disease. A prospective single blind randomized controlled design was used. Newly diagnosed PD patients were randomly assigned to three treatment groups: Madopar monotherapy group (n = 50), senfrol monotherapy group (n = 50) and placebo group (n = 50). Objective to study the performance of temporal working memory in PD patients and reveal the dopaminergic mechanism of temporal working memory.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for PD patients: age 50-80 years old; Junior high school or above, able to read and sign informed consent; Primary PD has just been diagnosed, Hoehn Yahr grade 1-2.5, and has not received any drug or non drug treatment.

The inclusion criteria of healthy control group: age 50-80 years old; Junior high school or above, able to read and sign informed consent.

Exclusion Criteria:

* The exclusion criteria of PD patients group were confirmed as secondary PD; Mental retardation, dementia or depression; Other neuropsychiatric diseases (such as epilepsy, schizophrenia), cerebrovascular diseases (such as stroke) or brain trauma; Antidepressants were used; History of alcohol dependence or drug abuse; Head MRI examination (such as claustrophobia, implantable medical device) is not allowed.

Exclusion criteria of healthy control group: Parkinson's disease symptoms (such as static tremor, bradykinesia, limb stiffness); Mental retardation, dementia or depression; REM sleep behavior disorder; There were symptoms of hypoosmia; Other neuropsychiatric diseases, cerebrovascular diseases or brain trauma; Antidepressants were used; History of alcohol dependence or drug abuse; No head MRI.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of cognition function | 12 months after the trail
  The score of MontrealCognitiveAssessment(MoCA),ranging from 0-30,with higher socre means better outcome

SECONDARY OUTCOMES:
Task state fMRI scanning | Before drug treatment
Task state fMRI scanning | 4 weeks after receiving drug treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yingshuang Zhang, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No